CLINICAL TRIAL: NCT04399941
Title: Role of Intravascular Ultrasound in Patients With End-stage Renal Disease on Dialysis
Brief Title: Intravascular Ultrasound in Patients With End-stage Renal Disease on Dialysis
Acronym: IVUS in ESRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-37396; 1R21DK119740-01A1 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: End Stage Renal Disease
Keywords: intravenous ultrasound (IVUS); central venous stenosis (CVS); hemodialysis; dialysis access malfunction; fistulogram; stenosis; virtual histology (VH-IVUS) software
MeSH Terms: conditions — Kidney Failure, Chronic; Constriction, Pathologic | interventions — Phlebography; Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IVUS and venography group (Experimental): Participants in the this group will receive venography/fistulogram, intravascular ultrasound (IVUS), and image processing.
  Interventions: Diagnostic Test: Venography; Diagnostic Test: Intravascular ultrasound (IVUS); Other: Image processing

INTERVENTIONS:
Diagnostic Test: Venography — The venography will be performed as part of the patient's standard of care. The dialysis access will be punctured upstream of the arteriovenous anastomosis in AVF or AVG using a 4-F coaxial access set (Micro- puncture; Cook, Inc, Bloomington, Indiana). The contrast will be injected intravenously by a pump with 200 psi and a bolus of 2m/sec for total of 5 ml during upper extremity vein filming and 10 ml of contrast bolus by 3 ml/s during central vein filming while holding the breath in inspiration in anterioposterior plane.
  Other Names: Fistulogram
Diagnostic Test: Intravascular ultrasound (IVUS) — IVUS will be performed through the same sheath of the coaxial access set using an Eagle Eye Platinum RX digital catheter 7F over a compatible guidewire under fluoroscopic guidance. The lesion will be estimated fluoroscopically from the marker IVUS catheter in the vein and the cranial and caudal margins of stenotic lesion will be directly visualized during pullback of the IVUS catheter.
Other: Image processing — Image processing will be performed by two radiologists in a blinded manner on the images devoid of personal identifier. An adjudication committee will oversee the process and confirm their findings in case of a discrepancy.

SUMMARY:
Hemodialysis represents a life line of patients with end stage renal disease, who are commonly maintained on hemodialysis through catheters. Prolonged exposure to these catheters eventually damages the walls of veins, which results in stenosis at the local site. This condition is called central venous stenosis (CVS) and affects number of patients on hemodialysis in the United States and can compromise the dialysis efficacy. The current diagnostic modality for CVS is venography, which has several limitations. This study proposes to examine intravenous ultrasound (IVUS) as a potentially superior modality, which will provide additional information.

ELIGIBILITY:
Inclusion Criteria:

* ESRD (end stage renal disease) patients at BMC (Boston Medical Center)
* Receiving hemodialysis
* Has a dialysis access malfunction
* Undergoing a diagnostic fistulogram for the dialysis access malfunction

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Extent of stenosis | 18 months
  The severity of venous stenosis will be assessed using venogram and IVUS results. It will be calculated as the percentage diameter or area reduction, expressed as the ratio of the MLD or MLA to the RVD or RVA.
Length of lesions | 18 months
  The length of each lesion will be measured between points with >50% diameter reduction in comparison to the referenced vein diameter and the referenced vein area at the pre-stenotic venous segment.
Morphology of lesion | 18 months
  The morphology of lesion will be defined as fibrotic and fibrofatty based on IVUS images.

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Chitalia, MD PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No